CLINICAL TRIAL: NCT05092841
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase III Study to Assess the Efficacy and Safety of PXT3003 in Charcot-Marie-Tooth Type 1A (CMT1A) Treated 15 Months
Brief Title: A Study to Assess the Efficacy and Safety of PXT3003 in Charcot-Marie-Tooth Type 1A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly GeneNet Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Tasly Pharmaceutical Group Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-CM-PXT3003-Ⅲ
Record Dates: First submitted 2021-09-26; First posted 2021-10-26 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Charcot-Marie-Tooth Type 1A
MeSH Terms: interventions — Naltrexone; Sorbitol; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PXT3003 (Experimental): Liquid oral solution, 10 mL twice a day, morning and evening with food
  Interventions: Drug: PXT3003
- PXT3003 Placebo (Placebo Comparator): Liquid oral solution, 10 mL twice a day, morning and evening with food
  Interventions: Drug: PXT3003 placebo

INTERVENTIONS:
Drug: PXT3003 — Patients will be administered PXT3003 twice daily (bid) at 10mL.
  Other Names: (RS)-baclofen, naltrexone hydrochloride and D-sorbitol oral fixed dose combination
  Arms: PXT3003
Drug: PXT3003 placebo — Patients will be administered PXT3003 placebo twice daily (bid) at 10mL.
  Other Names: liquid oral solution
  Arms: PXT3003 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled and multicenter 3 phase trial evaluating the therapeutic effect and safety of CMT1A by PXT3003. This double-blind study will assess in parallel groups 1 dose of PXT3003 compared to Placebo in CMT1A patients treated for 15 months.

DETAILED DESCRIPTION:
This multi-center, randomized, double-blind, placebo-controlled, Phase III clinical study is designed to evaluate PXT3003 versus placebo in subjects with genetically confirmed CMT1A of mild-to-moderate severity (CMTNS-V2 score >2 and ≤18) aged 16 to 65 years.

Genetically confirmed CMT1A subjects will be screened and randomized in a 1:1 ratio to receive either oral PXT3003 daily or matching placebo for 15 months. A total of approximately 176 subjects will be enrolled.

Visits will take place at Screening (up to -30 days), Baseline , and Months 3, 6, 9, 12, and 15.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 to 65 years (included boundary value), of either sex;
2. Patients with CMT1A (PMP22 duplication on chromosome 17p11.2) confirmed by gene diagnosis; 3.2 < CMTNS-v2 score ≤ 18;

4.Patients are dorsalis pedis flexor weakness at least (clinical evaluation); 5.Ulnar nerve motor nerve conductance velocity > 15 m/s; 6.Subjects participate in clinical trials and sign informed consent voluntarily , and they have the ability to understand as will as abide by research procedures.

Exclusion Criteria:

1. Being allergic to RS-baclofen, naltrexone HCL, D-sorbitol or any component in pxt3003 excipients or having other serious prior allergic reaction;
2. Existence contraindications of baclofen, naltrexone or sorbitol, such as porphyria;
3. Any other associated cause of peripheral neuropathy such as diabetes mellitus (including diabetes history and glycosylated hemoglobin >6.5%)
4. Subjects with other neurological diseases affecting the evaluation of study treatment;
5. Patients with the score of ONLS score is 0;
6. A history of unstable medical diseases with clinically significant unstable medical diseases (unstable angina pectoris, tumor, blood disease, hepatitis or liver failure, renal failure, etc.) that may cause harm to the subjects participating in this study in the past 1 year;
7. Limb surgery had implemented within the first six months of randomization or will be planned before the completion of the clinical trial;
8. Hepatic or renal dysfunction:

   1. TBIL>1.5×ULN,ALT>3×ULN,AST>3×ULN;
   2. Cr>1.5×ULN;
9. Syphilis antibody and HIV antibody positive subjects;
10. Subjects with tumors indicated by chest radiograph or B-ultrasound;
11. Subjects with alcohol dependence in recent 3 months;
12. Females that are of childbearing potential, pregnant, or are breast-feeding;Subjects who are unable to use appropriate contraceptives during the trial;
13. Subjects with concomitant treatment 4 weeks before enrollment, including but not limited to baclofen, naltrexone, sorbitol, opioids, vitamin C, levothyroxine and potentially neurotoxic drugs (such as amiodarone and chloroquine);
14. Subjects unable to complete the follow-up of study;
15. Participated in another clinical trial and used the test drug within the last 30 days;
16. Different subjects from the same family and living in the same residence can only include one subject, so as to avoid treatment confusion, affect blind treatment and affect the interpretation of the research results;
17. Investigators affirm the compliance in a certain subject is poor or there are some other factors that are not suitable to participate in this clinical trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Overall Neuropathy Limitation Scale (ONLS) score | 15 months
  The primary efficacy endpoint will be the main effect of the studied treatment on the improvement of disability measured by the Overall Neuropathy Limitation Scale (ONLS) score, summarized at 15 months defined by: the change of the ONLS from baseline to the 15 months.ONLS is a disability scale that was derived and improved from the Overall Disability Sum Score to measure limitations in the everyday activities of the upper limbs (rated in 5 points) and the lower limbs (rated on 7 points) . The total score goes from 0 ( no disability) to 12 (maximum disability).

SECONDARY OUTCOMES:
Treatment responders rate of PXT3003; | 15 months
  Responders Rate to PXT3003 therapy defined as a patients improving on ONLS at end of treatment.
The sub-item of Arm and leg scores in Overall Neuropathy Limitation Scale (ONLS) | 15 months
  ONLS is a disability scale that was derived and improved from the Overall Disability Sum Score to measure limitations in the everyday activities of the upper limbs (rated in 5 points) and the lower limbs (rated on 7 points) . The total score goes from 0 ( no disability) to 12 (maximum disability).
Total and sub-item score of Charcot-Marie-Tooth neuropathy score second version (CMTNS-V2); | 15 months
  CMTNS is a specific scale designed to assess severity of impairment in CMT disease .Although not completely validated, it provides a single and reliable measure of CMT severity. It is a 36-point scale based on 9 items: 5 of them quantify impairment (sensory symptoms, pin sensibility, vibration, arm and leg strength).
10-Meter Walk Test (10MWT); | 15 months
  Record the time for walk 10 meters . 10m WT is simple to administer, standardized, reliable and valid evaluation of functional exercise capacity and gait that has been proven reliable in neurologic disorders and in CMT patients. Results recorded are the time to walk 10 meters and the number of steps performed.
Nine-hole peg test (9HPT) for non-dominant hand ; | 15 months
  The 9-HPT is a simple timed test of fine motor coordination of extremities in the upper limbs.
Quantified Muscular Testing (QMT) (grip strength and bilateral foot dorsiflexion dynamometry) ; | 15 months
  QMT is used to evaluate motor strength in CMT1A. The following muscles will be evaluated: hand grip (right and left).
Electrophysiological parameters Sensory responses measured at ulnar and radial nerves on the non-dominant side: | 15 months
  The assessment parameters including: Distal motor latency (DML) .
Electrophysiological parameters motor responses measured at ulnar and radial nerves on the non-dominant side | 15 months
  The assessment parameters including: Nerve conduction velocity (NCV) .

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Director — Tasly Group,Co.Ltd.
Locations (25):
- China (25):
  - Peking University Third Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Nanfang Hospital Southern Medical University, Guangzhou
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Inner Mongolia People's Hospital, Hohhot
  - Qilu Hospital of Shandong University, Jinan
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Qilu Hospital of Shandong University（Qingdao）, Qingdao
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Renmin Hospital of Wuhan University（Hubei General Hospital）, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No